CLINICAL TRIAL: NCT06742788
Title: The Feasibility of Transcutaneous Auricular Vagus Nerve Stimulation on Pregnancy Outcomes of Infertility Patients Undergoing in Vitro Fertilization: Study Protocol for a Pilot Randomized Controlled Trial
Brief Title: The Feasibility of taVNS on Pregnancy Outcomes of Infertility Patients Undergoing IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Yonghong, MD, Associate Director of Neurology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20242351liuyonghong
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Infertility Assisted Reproductive Technology
Keywords: Infertility; Assisted Reproductive Techniques; Transcutaneous Auricular Vagus Nerve Stimulation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- the taVNS group (Experimental): The taVNS group receives Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) along with In Vitro Fertilization (IVF) treatment. The taVNS protocol is configured with a pulse width of 500 µs, a frequency of 25 Hz, and a current intensity titrated to each patient's pain tolerance threshold (range: 0.5-2.0 mA). The stimulation is to be carried out for a total of 1.5 hours daily, with the sessions divided into three parts, each lasting 30 minutes. At least one of these periods occur within 2 hours before bedtime.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)
- the staVNS group (Sham Comparator): The staVNS group receives sham transcutaneous auricular vagus nerve stimulation, along with In Vitro Fertilization (IVF) treatment. The staVNS protocol is set at a pulse width of 500 µs and a frequency of 25 Hz, with an intensity value of 0.1 mA.The stimulation of 0.1 mA acts as a therapeutic signal below the threshold level and functions as a sham stimulus. The stimulation is to be carried out for a total of 1.5 hours daily, with the sessions divided into three parts, each lasting 30 minutes. At least one of these periods occur within 2 hours before bedtime.
  Interventions: Device: sham transcutaneous auricular vagus nerve stimulation (staVNS)
- the IVF control group (No Intervention): The IVF control group refers to receiving only in vitro fertilization (IVF) treatment without any additional Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) treatment.

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) is an emerging, non-invasive adjunctive therapy.
  The taVNS protocol is configured with a pulse width of 500 µs, a frequency of 25 Hz, and a current intensity titrated to each patient's pain tolerance threshold (range: 0.5-2.0 mA). The stimulation is to be carried out for a total of 1.5 hours daily, with the sessions divided into three parts, each lasting 30 minutes. At least one of these periods occur within 2 hours before bedtime.
  The study will use the Chinese National Institutes for Food and Drug Control certificated taVNS device TVNS-100 (Xinzhile Medical Technology Co., Jiangxi, China). The study includes an intervening period of 4 weeks.
  Arms: the taVNS group
Device: sham transcutaneous auricular vagus nerve stimulation (staVNS) — The sham transcutaneous auricular vagus nerve stimulation (staVNS) serves as a sub-threshold therapeutic stimulus functions as a sham stimulus. The staVNS protocol is set at a pulse width of 500 µs and a frequency of 25 Hz, with an intensity value of 0.1 mA. The stimulation is to be carried out for a total of 1.5 hours daily, with the sessions divided into three parts, each lasting 30 minutes. At least one of these periods occur within 2 hours before bedtime. The study will use the Chinese National Institutes for Food and Drug Control certificated taVNS device TVNS-100 (Xinzhile Medical Technology Co., Jiangxi, China). The study includes an intervening period of 4 weeks.
  Arms: the staVNS group

SUMMARY:
To assess the feasibility of taVNS on pregnancy outcomes of infertility subjects undergoing IVF, the primary aim of this trial will focus on encompassing recruitment, compliance, and preliminary engagement outcomes.

The exploratory aim is to carry out clinical research, which entails evaluating the preliminary effects of the intervention in order to ascertain its potential benefits.

The main question it aims to answer is: Does the taVNS is feasible and tolerated in the context of IVF?

What medical problems do participants have when using the taVNS device? Researchers will compare the taVNS to the sham transcutaneous auricular vagus nerve stimulation (a look-alike device that produces a sub-threshold therapeutic stimulus and functions as a sham stimulus) and blank control to see if the taVNS device works to enhance outcomes of IVF.

Participants will:

Use the device a total of 1.5 hours daily, with the sessions divided into three parts, each lasting 30 minutes. At least one of these periods occur within 2 hours before bedtime.

Visit the clinic according to the scheduled treatment time points of IVF. Keep a diary of their adverse events and the number of times they use the device.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 20 to 40 years, diagnosed with infertility, and preparing to undergo IVF treatment;
2. Female subjects with anti-Müllerian hormone (AMH) > 1.2 ng/mL;
3. Scoring at mild-to-moderate levels of impairment on anxiety, and depression scales;
4. Both the subject and their family sign the informed consent form.

Exclusion Criteria:

1. The subject had been treated with taVNS in the past;
2. Subjects preparing to undergo frozen embryo transfer;
3. Subjects with a history of mental disorder or who score at a severe level of impairment on anxiety and depression scales;
4. Taking sedatives, anxiety, depression, or psychiatric medications;
5. Comorbidities including arrhythmia, hypertension, diabetes, chronic heart and kidney diseases;
6. Ineligibility for enrollment assessed by a gynecologist or neurologist;
7. Metallic implants or devices contraindicating taVNS.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the recruitment rate | The time frame for the recruitment rate is 12 months after the intervention begins.
  The recruitment rate refers to the number of eligible individuals screened.
the enrollment rate | The time frame for the enrollment rate is 12 months after the intervention begins.
  The the enrollment rate refers to the proportion of eligible patients who consent to participate.
the retention rate | The time frame for the retention rate spans from baseline to 4 weeks after ET.
  The retention rate refers to the proportion of enrolled individuals who do not withdraw from the intervention.
the patient adherence | The time frame for patient adherence spans from baseline to 4 weeks after ET.
  The patient adherence refers to the proportion of patients who complete the intervention.

SECONDARY OUTCOMES:
the total number of oocytes retrieved | On the day of oocyte retrieval
high-quality embryo rate | On the day of embryo transfer (day 14)
the positive rate of hCG | The positive rate of hCG will also be observed two weeks after ET
  The hCG level, specifically defined as >10 mIU/mL, is an important indicator of pregnancy success.
Clinical Pregnancy Rate | The primary efficacy outcome of the study is to measure and compare the difference in CPR among three groups 4 weeks after ET.
  Description: The clinical pregnancy rate (CPR) is a measure used in reproductive medicine to evaluate the success of in vitro fertilization (IVF) treatment. It is defined as the percentage of women who achieve a clinical pregnancy from the first fresh or frozen embryo transfer cycle. A clinical pregnancy is confirmed by ultrasound and is characterized by the presence of a gestational sac within the uterine cavity, as observed 4 weeks after the embryo transfer has taken place.
The Fertility Quality of Life Scale (FertiQoL, Simplified Chinese version) | The scale will be observed at baseline, the day of embryo transfer (day 14) and 2 weeks after embryo transfer.
  The Fertility Quality of Life Scale yields six subscale and three total scores with a range of 0 to 100. Higher scores mean higher quality of life and a better outcome.
Pittsburgh Sleep Quality Index (PSQI) | The scale and questionnaire measurement will be observed at baseline, the day of embryo transfer (day 14) and 2 weeks after embryo transfer.
  The total score range of the Pittsburgh Sleep Quality Index (PSQI) is from 0 to 21. Higher scores mean poorer sleep quality and a worse outcome.
14-item Hamilton Anxiety Rating Scale (HAMA-14) | The scale and questionnaire measurement will be observed at baseline, the day of embryo transfer (day 14) and 2 weeks after embryo transfer.
  The total score range of the 14-item Hamilton Anxiety Rating Scale (HAMA-14) is from 0 to 56. Higher scores mean more severe anxiety and a worse outcome.
17-item Hamilton Depression Rating Scale (HAMD-17) | The scale and questionnaire measurement will be observed at baseline, the day of embryo transfer (day 14) and 2 weeks after embryo transfer.
  The total score range of the 17-item Hamilton Depression Rating Scale (HAMD-17) is from 0 to 68. Higher scores mean more severe depression and a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Liu, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No